CLINICAL TRIAL: NCT03101488
Title: A Phase I, Single Arm, Multiple Dose, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability and Pharmacokinetics of KN035 Administered in Subcutaneous Injection as a Single Agent to Subjects With Advanced Solid Tumors
Brief Title: Phase I Study of KN035 in Chinese Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 3D Medicines (Sichuan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: 3D Medicines (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN035-CN-001
Record Dates: First submitted 2017-03-27; First posted 2017-04-05 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Solid Tumors
Keywords: KN035; phase 1
MeSH Terms: interventions — envafolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KN035 (Experimental): KN035 is to be injected subcutaneously 0.1mg/kg or 0.3mg/kg or 1mg/kg or 2.5mg/kg or 5mg/kg or 10mg/kg weekly until disease progresses or unacceptable tolerability occurs.
  Interventions: Drug: KN035

INTERVENTIONS:
Drug: KN035 — KN035 is a monoclonal antibody drug which is formulated for subcutaneous injection in a single-use vial (brown neutral borosilicate) containing a total of 300 mg antibody in 1.5 ml of solution.

SUMMARY:
This dose escalation and dose expansion study is to evaluate and characterize the tolerability and safety profile of single agent KN035 in Chinese adult subjects with unresectable advanced carcinoma.

DETAILED DESCRIPTION:
Dose escalation study is to evaluate the safety and tolerability of KN035 in advanced and metastatic solid tumor. Six dose levels are planned and include: 0.1, 0.3, 1.0, 2.5, 5, 10 mg/kg/dose. Subjects will be assigned to a dose level in the order of study entry. The first cohort of 1 subject will receive KN035 at 0.1 mg/kg/dose as a subcutaneous (sc) injection every week for a total of 4 injections (Days 1, 8, 15 and 22) in the first 28-day cycle. For the first 2 cohorts (0.1 and 0.3 mg/kg/dose), only one subject will be enrolled in each cohort until 1 subject experiences a ≥ Grade 2 drug-related adverse event in the first cycle, then 2 additional subjects will be enrolled at this cohort. Thereafter, the study will become the traditional 3+3 design with 3 or 6 subjects treated at this dose level and all subsequent dose levels depending upon the incidence of DLTs. However, if no ≥ Grade 2 drug-related adverse event occurs in the first 2 cohorts, starting with cohort 3, the study will become the traditional 3+3 design with 3 or 6 subjects enrolled.

Dose expansion-1 study is planned to conduct in advanced hepatocellular cancer subjects at 2.5 mg/kg and 5 mg/kg dose level, respectively.

Dose expansion-2 study is planned to conduct in advanced solid tumor subjects at 2.5 mg/kg and 5 mg/kg dose level, respectively

ELIGIBILITY:
Main Inclusion Criteria for dose escalation study:

* Subject is male or female ≥ 18 years and ≤ 70 years of age on the day of signing informed consent,and subject has voluntarily agreed to participate by giving written informed consent.
* Subjects must have a histopathological diagnosis of any locally advanced or metastatic solid tumor, Subjects must have failed established standard medical anti-cancer therapies ( have disease progression after the therapies or be intolerant to the therapies) or Subjects refuse to standard therapies, or no effective treatment.
* Measurable disease as defined by RECIST v1.1.
* Subject must have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Life expectancy ≥ 12 weeks.
* Subject must have adequate hematologic and organ function.
* Female subject of childbearing potential has a negative serum pregnancy test.
* Female subjects of childbearing potential and male subjects with partner of childbearing potential should agree to keep abstinence (refuse to heterosexual intercourse) or use one or more methods of contraception of which the failure rate is less than 1% per year starting with the first dose of study drug through at least 6 months after the last dose of study therapy.

Main Inclusion Criteria for dose expansion study:

* Histologic confirmation of advanced hepatocellular carcinoma, disease not eligible for curative surgical and/or locoregional therapies, OR progressive disease after surgical and /or locoregional therapies.
* At least one RECIST 1.1 measurable untreated lesion. All subjects must have at least one previously untreated, unidimensionally measurable lesion by contrast-enhanced spiral computed tomography (CT) ≥10 mm or contrast enhanced dynamic magnetic resonance imaging (MRI) scan ≥10 mm (malignant lymph nodes must be ≥15 mm on short axis).
* Subject is male or female ≥ 18 years and ≤ 75 years of age on the day of signing informed consent,and subject has voluntarily agreed to participate by giving written informed consent.
* Subject must have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Cirrhotic status of Child-Pugh Class A.
* Subjects are eligible to enroll if they have non-viral-HCC, or if they have HBV-HCC, or HCV-HCC defined as follows:

  i) HBV-HCC: Resolved HBV infection (as evidenced by detectable HBV surface antibody, detectable HBV core antibody, undetectable HBV DNA, and undetectable HBV surface antigen) or Chronic HBV infection (as evidenced by detectable HBV surface antigen or HBV DNA). Subjects with chronic HBV infection must have HBV DNA < 104 copies/ml and must be on antiviral therapy.

ii) HCV-HCC: Active or resolved HCV infection as evidenced by detectable HCV RNA or antibody.

* Life expectancy ≥ 12 weeks.
* Subject must have adequate hematologic and organ function.

Main Exclusion Criteria:

* Subject Is currently participating and receiving study therapy or has participated in a study of an investigational agent and receive study therapy within 28 days of the first dose of study drug.
* Subject has not recovered to CTCAE Grade 1 or better from the adverse events due to cancer therapeutics administered
* Subject has a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds (ms)), or a history of additional risk factors for torsade de pointes (TdP, e.g., heart failure, hypokalemia, family history of Long QT Syndrome), or is using concomitant medications that prolong the QT/QTc interval.
* Subject has had antineoplastic therapy within 4 weeks prior to the first dose of study therapy KN035.
* Subject is, with one year of the time signing informed consent, a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
* Subjects with symptomatic ascites, pleural effusion or pericardial effusion.
* Subject is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Subject has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to study entry, have no evidence of new or enlarging brain metastases and are off steroids for at least 7 days from first dose of KN035.
* Subject has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Subject has Leptomeningeal disease.
* Subject previously had a severe hypersensitivity reaction to treatment with another mAb.
* Subject has an active infection (CTCAE≥Grade 2) with 4 weeks of the first dose.
* Subject is positive for Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), active hepatitis B (HBV surface antigen positive and HBV DNA ≥ 104 copies/ml)or hepatitis C or tuberculosis (HCV antibody positive and HCV-RNA≥ 103 copies/ml).
* Subject has received or will receive a live vaccine within 4 weeks prior to the first administration of study drug.

Addtional exclusion criteria for dose expansion study:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* The patient accepted any anti-cancer therapy within 28 days prior to the first dose of study drug including surgery, radiotherapy, biotherapy, immunotherapy and/or locoregional therapy (eg: radiofrequency ablation [RFA], percutaneous ethanol [PEI] or acetic acid injection [PAI], cryoablation, high-intensity focused ultrasound [HIFU], transarterial chemoembolization [TACE], transarterial embolization [TAE], etc.)
* Prior liver transplant or history of hepatic encephalopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) in dose escalation study | From screening to up to cycle 1 (28 days)
Percentage of participants with adverse events (AEs), serious adverse events and AEs of special interest | From screening to up to 1 months after the last dose of study drug (up to approximately 2 years)
ORR of HCC patients in dose expansion study | Up to 2 approximately years

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of KN035 in Chinese patients | From Pre-dose of the first dose to up to cycle 12
Peak Time (Tmax) of KN035 in Chinese patients | From Pre-dose of the first dose to up to cycle 12
Area under the plasma concentration versus time curve (AUC) of KN035 in Chinese patients | From Pre-dose of the first dose to up to cycle 12
t1/2 of KN035 in Chinese patients | From Pre-dose of the first dose to up to cycle 12
Trough concentration of KN035 in Chinese patients | From Pre-dose of the first dose to up to cycle 12
Plasma clearance (CL) of KN035 in Chinese patients | From Pre-dose of the first dose to up to cycle 12
Apparent volume of distribution of KN035 in Chinese patients | From Pre-dose of the first dose to up to cycle 12
Accumulation rate of KN035 in Chinese patients | From Pre-dose of the first dose to up to cycle 12
Anti-Drug Antibody of KN035 in Chinese patients | From Pre-dose of the first dose to up to cycle 12
Changes of lymphocyte Subtyping | From Pre-dose of the first dose to up to cycle 12
Changes of cytokine | From Pre-dose of the first dose to up to 6 months
Objective Response Rate (ORR) | Up to 2 approximately years
Disease Control Rate (DCR) | Up to 2 approximately years
Progression-Free survival (PFS) | Up to 2 approximately years
Duration of Response (DOR) | Up to 2 approximately years
Correlation of tumor response with the PD-L1 expression | Up to 2 approximately years
Correlation of the tumor response with the expression of specific gene mutation | Up to 2 approximately years
overall survival | Up to 2 approximately years

CONTACTS AND LOCATIONS:
Overall Officials: jianming xu, Principal Investigator — Affiliated Hospital of Military academy of medical sciences
Locations (4):
- China (4):
  - Hunan Cancer Hospital, Changsha, Hunan
  - First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Affiliated Hospital of Military academy of medical sciences, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cui C, Wang J, Wang C, Xu T, Qin L, Xiao S, Gong J, Song L, Liu D. Model-informed drug development of envafolimab, a subcutaneously injectable PD-L1 antibody, in patients with advanced solid tumors. Oncologist. 2024 Sep 6;29(9):e1189-e1200. doi: 10.1093/oncolo/oyae102. PMID 38982653